CLINICAL TRIAL: NCT03266497
Title: Diet Quality Among U.S.-Born and Foreign-born Non-Hispanic Blacks: NHANES 2003-2012 Data
Brief Title: Diet Quality Among U.S.-Born and Foreign-born Non-Hispanic Blacks
Status: Completed | Type: Observational
Sponsor: Sara C. Folta (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Sara C. Folta, Associate Professor, Tufts University
Organization: Tufts University (Other)
Other Study IDs: R01HL115189 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Diet Habit
Keywords: diet quality; health disparities; immigrants; foreign-born; Blacks/African Americans; place of birth/nativity; length of residency; NHANES; acculturation
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study compares the diet quality between U.S.-born and foreign-born non-Hispanic Blacks using pooled NHANES data.

DETAILED DESCRIPTION:
This study uses the Alternative Healthy Eating Index-2010 (AHEI-2010) and Dietary Approach to Stop Hypertension (DASH) scores to compare diet quality between U.S.-born (n=3,837) and foreign-born (n=406) non-Hispanic Black adults aged 22-79y, based on pooled nationally representative data (NHANES 2003-2012); as well as by length of U.S. residency. Association between nativity and diet quality was done using multivariable-adjusted linear regression for the continuous total diet quality scores and their components, or multinomial (polytomous) logistic regression for categorical tertiles (low, medium, or high) of the total scores and their components. The study found that foreign-born Blacks had significantly higher AHEI-2010 and DASH scores compared to U.S-born Blacks, and more favorable intakes for many of the score components. Among foreign-born Blacks, diet quality did not significantly differ by length of residency. Foreign-born Blacks were more likely to be in the high than low tertile for fruit (including and excluding fruit juice), vegetables (excluding starchy vegetables), percent whole grains, and omega-3 fatty acids. Overall, the study suggests that foreign-born Blacks have better diet quality compared to their U.S.-born counterparts. Considering nativity among U.S. Blacks in nutrition research and public health efforts may therefore improve accuracy of characterizing dietary intakes and facilitate development of targeted nutrition interventions to reduce diet-related diseases in the diverse Black population in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* 22-79

Exclusion Criteria:

* Pregnant subjects
* Energy intakes of ≤600 kcal and ≥ 4800 kcal
* No dietary data available

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprised 4,243 non-Hispanic Blacks, including 3,837 U.S.-born (90.4%) and 406 foreign-born (9.6%). Compared to U.S.-born Blacks, a higher proportion of foreign-born Blacks were male, had attained a higher level of education, were classified as normal or overweight, had never been a smoker, engaged in physical activity, and had lower energy intake. In comparison to those who were in the U.S. for <10 years, more foreign-born Blacks who were in the U.S. for ≥30 years were current smokers (14.8% vs. 5.0%, respectively), had higher income (IPR of ≥4.00: 43.5% vs 7.9%, respectively), and a higher percent with a college degree or higher (39.4% vs. 18.3%, respectively). Foreign-born Blacks residing in the U.S. for ≥30 years reported higher BMI in comparison to those residing in the U.S. for <10 years (28.8 vs. 26.7 kg/m2).
Sampling Method: Probability Sample
Enrollment: 4243 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adapted AHEI-2010 | 2003-2012
  Components include: fruit (excluding fruit juice) (s/d); vegetables (excluding white potatoes) (s/d); whole grains (oz-equivalents/d); sugar-sweetened beverages (s/d); nuts, legumes, and vegetable protein (oz-equivalents/d); red/processed meat (s/d); long-chain omega-3 fats (EPA+DHA; mg/d); polyunsaturated fats (PUFA; % kcal/d); sodium (mg/d); and alcohol (drinks/d). Potential range of 0-100 points and higher scores indicative of higher diet quality

SECONDARY OUTCOMES:
Adapted DASH score | 2003-2012
  Quintile-, food-based dietary score assessing adherence to the DASH diet, which was developed as a dietary approach to prevent and treat hypertension. Components of the revised score include vegetables, fruit, whole grains, nuts and legumes, sodium, red and processed meat, and sugar-sweetened beverages.

IPD SHARING:
Plan to Share IPD: No